CLINICAL TRIAL: NCT02360592
Title: Combination Therapy of Interferon Alfa-2b Plus Interleukin 2 and Hepatitis B Vaccine in Entecavir-experienced Chronic Hepatitis B Patients With HBeAg Seroclearance: a Prospective, Randomized Open-label Trial (Endeavor Study, a Pilot Study)
Brief Title: Combination Therapy With Interferon Plus Interleukin 2 and Hepatitis B Vaccine in Chronic Hepatitis B Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: Beijing Kawin Technology Share-Holding Co., Ltd. (Industry); Fujian Cosunter Pharmaceutical Co. Ltd (Industry)
Responsible Party: Principal Investigator, Qin Ning, Director and Chair of Department of Infectious Diseases, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endeavor study, a pilot study
Record Dates: First submitted 2015-02-02; First posted 2015-02-10 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis B, Chronic
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — entecavir; Interferon alpha-2; Interleukin-2; Hepatitis B Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1, conventional control group (Active Comparator): Entecavir 0.5 mg po daily for 72 weeks
  Interventions: Drug: Entecavir
- 2, combination and sequential group (Experimental): Interferon alfa-2b 600wIU qod iH for 48 weeks plus Entecavir 0.5mg qd po for 8 weeks
  Interventions: Drug: Entecavir; Drug: Interferon alfa-2b
- 3, multitarget group (Experimental): Interferon alfa-2b 600wIU qod iH for 48 weeks plus Entecavir 0.5mg qd po for 8 weeks plus interleukin 2 25 wIU qod iH for 12 weeks plus Hepatitis B Vaccine 60ug qm im for 48 weeks
  Interventions: Drug: Entecavir; Drug: Interferon alfa-2b; Drug: Interleukin 2; Drug: Hepatitis B Vaccine

INTERVENTIONS:
Drug: Entecavir — In arm 1, Entecavir is used for 48 weeks and the follow up 24 weeks as conventional control, In arm 2 and 3, Entecavir is used for 8 weeks.
  Other Names: ETV
Drug: Interferon alfa-2b — In arm 2 and 3, interferon alfa-2b is used for 48 weeks
  Other Names: IFN a-2b
  Arms: 2, combination and sequential group; 3, multitarget group
Drug: Interleukin 2 — In arm 3, Interleukin 2 is used for 12 weeks
  Other Names: IL-2
  Arms: 3, multitarget group
Drug: Hepatitis B Vaccine — In arm 3, Hepatitis B Vaccine is used for 48 weeks
  Arms: 3, multitarget group

SUMMARY:
This study is a multi-center, randomized, prospective, open-label Phase IV Clinical trial to evaluate efficacy and safety of interferon alfa-2b therapy combinated with interleukin 2 and hepatitis B therapeutic vaccine versus interferon alfa-2b alone in chronic hepatitis B patients with entecavir achieving HBeAg seroclearance. Patients were randomized to one of 3 groups to receive different antiviral treatment.

DETAILED DESCRIPTION:
Patients who have been pretreated with entecavir for at least one year, with HBV (Hepatitis B Virus) DNA less than 1000 copies/ml and HBeAg seroclearance were randomized to one of 3 groups, to receive Entecavir 0.5 mg po daily for 72 weeks, or Interferon alfa-2b 600wIU qod iH for 48 weeks plus Entecavir 0.5mg qd po for 8 weeks, or Interferon alfa-2b 600wIU qod iH for 48 weeks plus Entecavir 0.5mg qd po for 8 weeks plus interleukin 2 25 wIU qod iH for 12 weeks plus Hepatitis B Vaccine 60ug qm im for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients from 18 to 65 years of age;
2. Undergoing treatment with entecavir for at least 1 year ;
3. HBsAg(+), HBeAg(+), HBV DNA≥ 100000 copies/ml，ALT≥2 ULN and ≤10 ULN before receiving entecavir treatment;
4. HBV DNA ≤1000 copies/mL;
5. HBeAg (-);
6. HBsAg (+);
7. Negative urine or serum pregnancy test (for women of childbearing potential) documented within the 24-hour period prior to the first dose of test drug;
8. Liver biopsy confirmed without cirrhosis (optional);
9. Agree to participate in the study and sign the patient informed consent.

Exclusion Criteria:

1. Patients who had NAs resistance;
2. Other antiviral, anti-neoplastic or immunomodulatory treatment (including supra physiologic doses of steroids and radiation) 6 months prior to the first dose of randomized treatment (except for 7 days of acyclovir for herpetic lesions more than 1 month prior to first administration of randomized treatment). Patients who are expected to need systemic antiviral therapy other than that provided by the study at any time during their participation are also excluded;
3. Women with ongoing pregnancy or breast-feeding;
4. Co-infection with active hepatitis A, hepatitis C, hepatitis D(Those hospitals which have the ability to do the test will do) and/or human immunodeficiency virus (HIV);
5. ALT >10 ULN;
6. Evidence of decompensated liver disease (Child-Pugh score > 5 ). Child-Pugh > 5 means, if one of the following 6 conditions are met, the patient has to be excluded: a. Serum albumin < 3.5 g/L; b. Prothrombin time > 3 seconds prolonged; c. Serum bilirubin > 34 μ mol/L; d. History of encephalopathy; e. History of variceal bleeding; f. Ascites;
7. History or other evidence of a medical condition associated with chronic liver disease other than viral hepatitis (e.g., hemochromatosis, autoimmune hepatitis, metabolic liver disease, alcoholic liver disease, toxin exposures, thalassemia);
8. Signs or symptoms of hepatocellular carcinoma, patients with a value of alpha-fetoprotein > 100 ng/mL are excluded, unless stability (less than 10% increase) has been documented over at least the previous 3 months. Patients with values < 20 ng/mL but > 100 ng/mL may be enrolled, if hepatic neoplasia has been excluded by liver imaging;
9. Neutrophil count < 1500 cells/mm3 or platelet count <90,000 cells/mm3 at screening;
10. Hemoglobin < 11.5 g/dL for females and <12.5 g/dL for men;
11. Serum creatinine level > 1.5 ULN in screening period.
12. Phosphorus < 0.65 mmol/L;
13. ANA > 1:100;
14. History of severe psychiatric disease, especially depression. Severe psychiatric disease is defined as treatment with an antidepressant medication or a major tranquilizer at herapeutic doses for major depression or psychosis, respectively, for at least 3 months at any previous time or any history of the following: a suicidal attempt hospitalization for psychiatric disease, or a period of disability due to a psychiatric disease;
15. History of a severe seizure disorder or current anticonvulsant use;
16. History of immunologically mediated disease, (e.g., inflammatory bowel disease, idiopathic thrombocytopenic purpura, lupus erythematosus, autoimmune hemolytic anemia, scleroderma, rheumatoid arthritis etc.);
17. History of chronic pulmonary disease associated with functional limitation;
18. Diseases that IFN and Nucleotides or nucleosides are not suitable.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Percentage of HBsAg loss at week 48 | week 48
  Change from baseline in Percentage of HBsAg loss at week 48

SECONDARY OUTCOMES:
decline from baseline in HBsAg quantification at week 48 | week 48
  HBsAg quantification are measured.
Change from baseline in HBsAg seroconversion at week 48 | week 48
  HBsAg seroconversion from baseline is measured.

OTHER OUTCOMES:
Percentage of HBeAg seroconversion at week 48 | week 48
  Percentage of HBeAg seroconversion are measured at week 48
Percentage of HBV DNA normalization | week 48
  Percentage of HBV DNA normalization is measured.
Percentage of sustained virology response at week 72 | week 72
  Sustained virology response is measure at follow up week 24
Percentage of ALT normalization at week 48 | week 48
  Percentage of ALT normalization at week 48 is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Qin Ning, Ph.D. M.D., Principal Investigator — Department of Infectious Diseases, Tongji Hospital
Locations (12):
- China (12):
  - Anhui Provincial Hospital, Hefei, Anhui
  - BeiJing YouAn Hospital, Capital Medical University, Beijing, Beijing Municipality
  - First Hospital, Beijing University, Beijing, Beijing Municipality
  - People'S Hospital Under Beijing University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Department of infectious disease, Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Tongji Hospital, Wuhan, Hubei
  - Departmen of infectious disease, Xiangya Hospital, Central-south Universit, Changsha, Hunan
  - ShengJing Hospital of China Medical University, Shenyang, Liaoning
  - Shanghai Ruijin Hospital, Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital of College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The first affiliated hospital of Wenzhou medical universtiy, Wenzhou, Zhejiang